CLINICAL TRIAL: NCT01886638
Title: Determining the Effect of Abacavir on Platelet Activation in Virologically Suppressed HIV Positive Men: an Open Label Interventional Study
Brief Title: Determining the Effect of Abacavir on Platelet Activation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayside Health (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 248-13; ACTRN12613000570785 (Registry Identifier: ANZCTR)
Record Dates: First submitted 2013-06-24; First posted 2013-06-26 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: HIV; Cardiovascular Disease
Keywords: Platelets; HIV; Cardiovascular disease; Acute myocardial infarction; Abacavir; Antiretrovirals
MeSH Terms: conditions — Cardiovascular Diseases | interventions — abacavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abacavir (Experimental): Abacavir 600mg (as two 300mg tablets) once daily for 15 days
  Interventions: Drug: Abacavir

INTERVENTIONS:
Drug: Abacavir
  Other Names: Ziagen

SUMMARY:
HIV positive patients have a two fold increased risk of developing cardiovascular disease (such as heart attacks and strokes). Cardiovascular disease appears to be due in part to both HIV and the side effects from anti-HIV medications.

Abacavir (an important component of current HIV treatment regimens) is one medication shown to be associated with an increase the risk of heart attacks in some studies. The mechanism by which abacavir does this is unknown.

We hypothesise that abacavir is leading to heart disease by interacting with platelets, which then form blood clots within the arteries supplying the heart, the subsequent blockage of the artery causing a heart attack.

This study aims to determine if abacavir increases the activity (or "stickiness") of platelets, and thus provide evidence as to how it may be promoting heart attacks.

It will consist of 23 HIV positive men who currently have well controlled HIV. Participants will take abacavir for 15 days in addition to their usual anti-HIV medications. A blood sample to assess platelet activity will be taken at baseline, following the 15 days of therapy (i.e. at the time of maximal abacavir effect) and again after a 28 day washout period (to determine if any effects are reversible).

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* Male
* HIV positive
* Stable non-abacavir containing anti-retroviral regimen
* Undetectable HIV Viral load

Exclusion Criteria:

* HLA-B*57*01 allele positivity
* Previous allergy to abacavir
* Known cardiovascular disease
* High Baseline cardiovascular risk (Framingham risk score > 20%)
* Current or recent antiplatelet therapy
* Pre-existing platelet or bleeding disorder (i.e. Thrombophilia, Thrombocytopenia, Von willebrands disease, Haemophilia)
* Significant Chronic liver disease
* Current Methadone use

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-08; Primary Completion 2014-06 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change in Phosphorylated Vasodilator Stimulated Phosphoprotein (P-VASP) assay | Baseline, day 15 and day 48

SECONDARY OUTCOMES:
Platelet aggregation | Baseline, Day 15 and day 48
  Measurement of the degree of platelet aggregation in response to collagen related peptide and thrombin receptor-agonist peptide
Platelet specific collagen receptor glycoprotein VI (GPVI) | Baseline, Day 15 and Day 48
  Measurement of the expression and shedding of platelet specific collagen receptor GPVI

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Hoy, MBBS FRACP, Principal Investigator — Alfred health, Monash University; Janine Trevillyan, MBBS FRACP, Principal Investigator — Alfred Health, Monash university
Locations (1):
- Alfred Health, Melbourne, Victoria, Australia